CLINICAL TRIAL: NCT05584462
Title: Prevalence Of Gastroparesis In Type2 Diabetic Patients In Assiut University Hospital And Value Of Nuclear Imaging In Diagnosis
Brief Title: Gastroparesis in type2 Diabetic Patient
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mena Adly Wahba Tous, Assistant Lecturer, Assiut University
Other Study IDs: diabetic gastroparesis
Record Dates: First submitted 2022-10-10; First posted 2022-10-18 (Actual); Last update posted 2023-01-17 (Actual); Status verified 2023-01

CONDITIONS: Diabetic Gastroparesis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Gastroparesis is defined by objective delaying of gastric emptying without any evidence of mechanical obstruction. Diabetic gastroparesis is a potential complication that occurs in the setting of poorly controlled diabetes, resulting from dysfunction in the coordination and function of the autonomic nervous system, neurons, and specialized pacemaker cells (interstitial cells of Cajal, ICC) of the stomach and intestine, and the smooth muscle cells of the gastrointestinal tract

DETAILED DESCRIPTION:
Hyperglycemia (random blood glucose greater than 200 mg/dL), commonly seen in uncontrolled diabetes, has been associated with diabetic gastroparesis resulting from neuropathy in the setting of chronic hyperglycemia and does not resolve with improved glycemic control. Acute hyperglycemia, on the other hand, though it can also result in delayed gastric emptying, is often reversible with improved glycemic control. Although there is a stronger association between type 1 diabetes and gastroparesis, the incidence of type 2 diabetes is much greater, and therefore, gastroparesis associated with type 2 diabetes is seen more frequently. Additionally, incretin mimetics are used to treat patients with type 2 diabetes, and these medications pose an additional risk factor for developing gastroparesis.Gastric emptying scintigraphy (GES) is the investigation of choice for evaluating the disorders of gastric emptying because it is a simple, physiological, and sensitive investigation to objectively assess gastric emptying. Standard imaging is performed at 0,1,2,4 hours postprandially. A four-hour study is more sensitive and accurate in diagnosing gastroparesis, and clinicians should avoid shortened 2- and 3-hour studies.

ELIGIBILITY:
Inclusion Criteria:

1. Type 2 DM
2. Age < 40 years
3. >5 years of DM

Exclusion Criteria:

1. Type 1 DM
2. History of GIT surgry
3. Medical disease affect gastric emptying
4. Using of prokinetic

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: type2 diabetic patient in assiut university hospital
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
prevalence of gastroparesis in type 2 diabetic patients | 3 years

SECONDARY OUTCOMES:
Value of nuclear imaging (Gastric emptying scintigraphy) in diagnosis of gastroparesis | 3 years
  using of Gastric emptying scintigraphy as a tool for diagnosis of gastroparesis

CONTACTS AND LOCATIONS:
Overall Officials: Manal Ez Eldin, Study Director — Assiut University; Marwa Abo kresha, Study Director — Assiut University; Waleed Ahmed Mohamed, Study Director — Assiut University; mena adly wahba, Principal Investigator — Assiut University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Fehnel S, Fiedorek FT, Nelson L, DiBenedetti D, Spence S, Carson RT. Development and psychometric evaluation of the Diabetic Gastroparesis Symptom Severity Diary. Clin Exp Gastroenterol. 2019 Feb 22;12:93-103. doi: 10.2147/CEG.S184016. eCollection 2019. PMID 30863134
- [Background] Chedid V, Halawi H, Brandler J, Burton D, Camilleri M. Gastric accommodation measurements by single photon emission computed tomography and two-dimensional scintigraphy in diabetic patients with upper gastrointestinal symptoms. Neurogastroenterol Motil. 2019 Jun;31(6):e13581. doi: 10.1111/nmo.13581. Epub 2019 Mar 13. PMID 30868676
- [Background] Parkman HP, Wilson LA, Hasler WL, McCallum RW, Sarosiek I, Koch KL, Abell TL, Schey R, Kuo B, Snape WJ, Nguyen L, Farrugia G, Grover M, Clarke J, Miriel L, Tonascia J, Hamilton F, Pasricha PJ. Abdominal Pain in Patients with Gastroparesis: Associations with Gastroparesis Symptoms, Etiology of Gastroparesis, Gastric Emptying, Somatization, and Quality of Life. Dig Dis Sci. 2019 Aug;64(8):2242-2255. doi: 10.1007/s10620-019-05522-9. Epub 2019 Mar 9. PMID 30852767
- [Background] Revicki DA, Speck RM, Lavoie S, Puelles J, Kuo B, Camilleri M, Almansa C, Parkman HP. The American neurogastroenterology and motility society gastroparesis cardinal symptom index-daily diary (ANMS GCSI-DD): Psychometric evaluation in patients with idiopathic or diabetic gastroparesis. Neurogastroenterol Motil. 2019 Apr;31(4):e13553. doi: 10.1111/nmo.13553. Epub 2019 Feb 7. PMID 30734412
- [Background] Abell TL, Kedar A, Stocker A, Beatty K, McElmurray L, Hughes M, Rashed H, Kennedy W, Wendelschafer-Crabb G, Yang X, Fraig M, Omer E, Miller E, Griswold M, Pinkston C. Gastroparesis syndromes: Response to electrical stimulation. Neurogastroenterol Motil. 2019 Mar;31(3):e13534. doi: 10.1111/nmo.13534. Epub 2019 Jan 31. PMID 30706646
- [Background] Moshiree B, Potter M, Talley NJ. Epidemiology and Pathophysiology of Gastroparesis. Gastrointest Endosc Clin N Am. 2019 Jan;29(1):1-14. doi: 10.1016/j.giec.2018.08.010. PMID 30396519